CLINICAL TRIAL: NCT00099320
Title: Safety and Efficacy of Exenatide in Patients With Type 2 Diabetes Using Thiazolidinediones or Thiazolidinediones and Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-MC-GWAP
Record Dates: First submitted 2004-12-10; First posted 2004-12-13 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide; exendin-4; diabetes; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): After a 2-week placebo lead-in period, exenatide will be given in an esclating dose along with the subject's current therapy regimen
  Interventions: Drug: exenatide
- Placebo (Placebo Comparator): After a 2-week placebo lead-in period, subjects will be given placebo (in equivalent amounts to exenatide) in addition to their current therapy regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: exenatide — After a 2-week placebo lead-in period (twice daily, given subcutaneously) in addition to their current therapy regimen, subjects will administer 20 mcg of exenatide (2 units [5 μg] ), twice daily by subcutaneous injection, for the first 4 weeks of therapy, and then 40 μL of study drug (4 units [10 μg] of exenatide) twice daily by subcutaneous injection, for the remaining 12 weeks of therapy.
  Other Names: Byetta; AC2993; synthetic exendin-4
  Arms: Exenatide
Drug: Placebo — After a 2-week placebo lead-in period (twice daily, given subcutaneously) in addition to their current therapy regimen, subjects will administer placebo (in equivalent amounts to exenatide) for 16 weeks of therapy.
  Arms: Placebo

SUMMARY:
This study is designed to compare the effects of twice-daily exenatide plus oral antidiabetic (OAD) agents and twice-daily placebo plus OAD with respect to glycemic control, as measured by hemoglobin A1c (HbA1c), in patients with type 2 diabetes who experience inadequate glycemic control with OAD alone.

ELIGIBILITY:
Inclusion Criteria:

* Treated with thiazolidinedione (TZD) alone or in combination with metformin. TZD dose stable for at least 120 days prior to screening, and those patients on metformin must have been on a stable dose for at least 30 days prior to screening.
* HbA1c between 7.1% and 10.0%, inclusive.
* Body mass index (BMI) between 25 kg/m^2 and 45 kg/m^2.

Exclusion Criteria:

* Patient previously in a study using exenatide or GLP-1 analogs.
* Treated with oral anti-diabetic medications other than TZD and metformin within 3 months of screening.
* Treated with oral insulin within 3 months of screening.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2004-05; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated hemoglobin) from Baseline to Week 16, and if measured, any visits in between | Baseline, Week 4, Week 8, Week 12, Week 16
  Change in HbA1c from Baseline (Visit 3) to study termination at Week 16, and at all study visits in between
Change from Baseline to Week 16 in fasting serum glucose (FSG) and glucose | Baseline, Week 16
  Change from Baseline to Week 16 in FSG and glucose measured at different times throughout the day derived from 7-point self-monitored glucose (SMG) profile (glucose measurements before and 2 hours after the start of the morning, midday, and evening meals, and at bedtime)

SECONDARY OUTCOMES:
Percentage of subjects reaching the target HbA1c (<7%) | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
  The percentage of subjects reaching the target HbA1c (<7%) will be summarized and compared by treatment
Change in body weight from Baseline to Week 16 | Baseline, Week 16
  Change in body weight (kg) from Baseline to Week 16
Change from Baseline to Week 16 in fasting serum glucose (FSG) and glucose | Baseline, Week 16
  Change from Baseline to Week 16 in FSG and glucose measured at different times throughout the day derived from 7-point self-monitored glucose (SMG) profile (glucose measurements before and 2 hours after the start of the morning, midday, and evening meals, and at bedtime)
Changes in beta cell function and insulin sensitivity between Baseline and Week 16 | Baseline, Week 16
  Changes in beta cell function and insulin sensitivity as assessed by homeostasis model assessment (HOMA) analyses and the proinsulin/insulin ratio Between Baseline and Week 16
Changes in lipids between Baseline and Week 16 | Baseline, Week 16
  Changes from Baseline to Week 16 in serum lipids (total cholesterol [TC], high-density lipoprotein cholesterol [HDL-C], fasting triglycerides, calculated low-density lipoprotein cholesterol [LDL-C]

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (51):
- United States (40):
  - Research Site, Birmingham, Alabama
  - Research Site, La Jolla, California
  - Research Site, San Mateo, California
  - Research Site, Santa Barbara, California
  - Research Site, Spring Valley, California
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Idaho Falls, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Kalamazoo, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Butte, Montana
  - Research Site, McCook, Nebraska
  - Research Site, North Platte, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Scottsbluff, Nebraska
  - Research Site, Princeton, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Greenville, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Georgetown, Texas
  - Research Site, San Antonio, Texas
  - Research Site, The Colony, Texas
  - Research Site, Olympia, Washington
  - Research Site, Renton, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Huntington, West Virginia
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Dartmouth, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Spain (5):
  - Research Site, Granada
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Zaragoza

REFERENCES:
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356
- [Derived] Zinman B, Hoogwerf BJ, Duran Garcia S, Milton DR, Giaconia JM, Kim DD, Trautmann ME, Brodows RG. The effect of adding exenatide to a thiazolidinedione in suboptimally controlled type 2 diabetes: a randomized trial. Ann Intern Med. 2007 Apr 3;146(7):477-85. doi: 10.7326/0003-4819-146-7-200704030-00003. PMID 17404349